CLINICAL TRIAL: NCT06218498
Title: Comparison of an Non-ablative Fractional 1565nm vs. an Ablative 2940-nm Fractional Erbium-glass Laser for the Treatment of Male Androgenetic Alopecia
Brief Title: Comparison of an Non-ablative Fractional 1565nm vs. an Ablative 2940-nm Fractional Er Laser for the Treatment of Androgenetic Alopecia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20230943
Record Dates: First submitted 2024-01-02; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2023-11

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia | interventions — Lasers, Solid-State; Minoxidil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ablative fractional 2940-nm erbium yttrium aluminum garnet (Er: YAG) laser (Experimental)
  Interventions: Device: ablative fractional 2940-nm Er: YAG laser
- non-ablative fractional 1565nm (Experimental)
  Interventions: Device: non-ablative fractional 1565nm
- 5% minoxidil (Active Comparator)
  Interventions: Drug: 5% Minoxidil

INTERVENTIONS:
Device: ablative fractional 2940-nm Er: YAG laser — Ablative fractional 2940-nm Er: YAG laser (Dermablate MCL31, Asclepion Laser Technologies, Germany), the following parameters were used: model of N25%, energy density of 20-30J/cm2, pulse time of 300μs and one to two passes.
  Arms: ablative fractional 2940-nm erbium yttrium aluminum garnet (Er: YAG) laser
Device: non-ablative fractional 1565nm — Non-ablative fractional 1565nm (Lumenis, M22): Resur Fx len, energy of 30-35J/cm2, density of 200spot/cm2, overlap ≤10%.
  Arms: non-ablative fractional 1565nm
Drug: 5% Minoxidil — topical 5% minoxidil, 1 ml, twice daily
  Arms: 5% minoxidil

SUMMARY:
Laser sources have established their potential effect in inducing hair regrowth. No study has compared the effect of ablative fractional 2940-nm erbium yttrium aluminum garnet (Er: YAG) laser and non-fractional 15650nm fractional laser in the treatment of androgenetic alopecia (AGA).

DETAILED DESCRIPTION:
The investigators performed a prospective study between to compare the efficacy and safety of ablative fractional 2940-nm erbium yttrium aluminum garnet (Er: YAG) laser and non-fractional 15650nm fractional laser in the treatment of androgenetic alopecia (AGA). The efficacy of the two therapies was evaluated by the investigator's Global Assessment (IGA) scores and the patient's Likert satisfaction scale at week 12 and week 24. Changes in total, terminal and villous hair count, total and terminal hair diameter, and AGA grade were also recorded. Adverse events were evaluated at each follow-up.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65 years;；
* clinical diagnosis of AGA；
* AGA diagnosis was evaluated following Norwood Hamilton grade II-V criteria；
* no previous laser treatments for AGA in the past six months before enrollment；
* willingness to provide pictures and follow-up studies.

Exclusion Criteria:

* if presented with severe diseases of internal organs, eyes, or skin;
* inflammation, infection, or unhealed wounds on the skin around the site of treatment on the head;
* systematic treatment with corticosteroids or other immunosuppressants and immunomodulators in the past 3 months

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2023-11-24 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
TAHC | week 24
  Use the trichoscopy to assess the changing number of non-vellus hairs in the target area .

SECONDARY OUTCOMES:
HGQA | week 8, week 12, week 16, week 24, week 36
  Hair growth questionnaire assessment
TAHC | week 8, week 12, week 20, week 36
  Use the trichoscopy to assess the changing number of non-vellus hairs in the target area
TAHW | week 8, week 12, week 16, week 24, week 36
  Use the trichoscopy to assess the changing diameter of non-vellus hairs in the target area
IGA | week 8, week 12, week 16, week 24, week 36
  Investigator's Global Assessment. IGA was evaluated using a 7-point scale as follows: -3= obvious reduction of hair; -2= moderate reduction of hair; -1= mild reduction of hair; 0= change; 1= mild growth of hair; 2= moderate growth of hair; 3= obvious growth of hair.
Grade of Norwood-Hamilton | week 12, week 24, week 36
  The Grade of Norwood-Hamilton Classification
SSA | week 8, week 12, week 16, week 24, week 36
  Subject self-assessment. SSA was evaluated using a 7-point scale as follows: -3= obvious reduction of hair; -2= moderate reduction of hair; -1= mild reduction of hair; 0= change; 1= mild growth of hair; 2= moderate growth of hair; 3= obvious growth of hair.

OTHER OUTCOMES:
Incidents of adverse events | through study completion, an average of 36 weeks
  Safety assessment

CONTACTS AND LOCATIONS:
Overall Officials: Xianjie Wu, Ph.D, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are not publicly available due to the privacy of research participants but are available from the sponsor upon reasonable request.